CLINICAL TRIAL: NCT02371785
Title: Robotic-Assisted Peripheral Intervention for Peripheral Arterial Disease
Acronym: RAPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-002
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Critical Limb Ischemia; Claudication; Percutaneous Vascular Intervention; Peripheral Vascular Intervention
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CorPath 200 System (Experimental): CorPath 200 System for remote delivery and manipulation of guidewires and balloon catheters during percutaneous vascular intervention.
  Interventions: Device: CorPath 200 System

INTERVENTIONS:
Device: CorPath 200 System — Remote delivery of guide wires and balloon catheters for use in percutaneous vascular interventions (PVI).

SUMMARY:
This study evaluates the performance of the CorPath 200 System to deliver guide wires and balloons to blockages in the arteries of the leg.

DETAILED DESCRIPTION:
The CorPath 200 System is currently marketed for remotely delivering guide wires, balloons and stents to blockages in the coronary arteries. This study will evaluate the feasibility of CorPath 200 System to deliver guide wires and balloons to blockages in non-coronary arteries.

Guide wires and balloons are delivered to blockages in the lower limbs manually by doctors.If this study shows that guide wires and balloons can be safely delivered to blockages in the lower limbs, then it will be an alternative for physicians.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion

  1. At least 18 years of age;
  2. Symptomatic disease: presence of critical limb ischemia (including tissue loss or rest pain), or lifestyle-limiting claudication requiring intervention in iliac and/or superficial femoral arteries;
  3. The subject or the legally authorized representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent.
* Angiographic Inclusion

Presence of superficial femoral artery and/or iliac stenosis (>50%) or occlusion of up to 50 mm in length as determined by angiogram prior to index interventional procedure.

Exclusion Criteria:

* General Exclusion

  1. Failure/inability/unwillingness to provide informed consent;
  2. Target vessel has been previously treated with bypass;
  3. Has an abdominal aortic aneurysm contiguous with the iliac artery target lesion;
  4. Has contraindication to anticoagulation;
  5. Has bleeding or a hypercoagulability disorder;
  6. Thrombocytopenia;
  7. Elevated international normalized ratio (>1.5);
  8. Elevated serum creatinine (≥2.5 mg/dL);
  9. Active infection;
  10. Contraindication to contrast; or
  11. Enrolled in concurrent clinical study.
* Angiographic Exclusion

  1. Target vessel:

     1. shows evidence of previous dissection or perforation, or
     2. has adjacent acute thrombus;
  2. Lesion is highly calcified;
  3. Lesion requires use of any atherectomy device during the procedure;
  4. Has a pre-existing target artery aneurysm or perforation or dissection of the target artery prior to initiation of the interventional procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2015-04-28 (Actual); Study Completion 2015-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Brodmann, M.D., Principal Investigator — Medizinische Universität Graz
Locations (1):
- Medizinische Univeristät Graz, Graz, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During February - April 2015 period 20 participants were enrolled in the RAPID study at one (1) clinical site.
Period: Overall Study
Arm/Group | CorPath 200 System
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Demographics: Baseline measures for the treated subjects.
Arm/Group | Baseline Demographics
Number analyzed (Participants) | 20
Age, Continuous [Median (Standard Deviation); unit: years] | 65.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Device Technical Success
Description: Number of lesions for which there was technical success" as accurate and appropriate.
Time Frame: Procedure
Population: 29 lesions treated in 20 subjects.
Measure: Number; unit: lesions
Units Other Than Participants: lesions
Arm/Group | CorPath 200 System
Number analyzed (Participants) | 20
Number analyzed (lesions) | 29
lesions | 29

2. Primary Outcome: Adverse Events
Description: No device-related serious adverse events during the procedure.
Time Frame: Procedure
Population: Device-related events that occured in subjects treated.
Measure: Count of Participants; unit: Participants
Groups:
- Device-related Periprocedural Event: The primary safety measure was the absence of device-related serious adverse events during the procedure. These were defined as adverse events related to the use of the robotic device that resulted in hospitalization, prolonged hospitalization, were life threatening, or resulted in death.
Arm/Group | Device-related Periprocedural Event
Number analyzed (Participants) | 20
Participants | 0

3. Secondary Outcome: Clinical Procedural Success
Description: Defined as <50% residual stenosis in all CorPath 200 System treated lesions at the completion of the interventional procedure (without an unplanned switch to the manual procedure) in the absence of device-related SAE, either within twenty-four (24) hours of the procedure or prior to hospital discharge, whichever occurs first.
Time Frame: 24-hours
Population: Achievement of <50% residual stenosis in all robotic system treated lesions at the completion of the interventional procedure without an unplanned switch to the manual procedure in the absence of device-related serious adverse events.
Measure: Number; unit: participants
Groups:
- Clinical Procedural Success: Defined as <50% residual stenosis in all CorPath 200 System treated lesions at the completion of the interventional procedure (without an unplanned switch to the manual procedure) in the absence of device-related SAE, either within twenty-four (24) hours of the procedure or prior to hospital discharge, whichever occurs first.
Arm/Group | Clinical Procedural Success
Number analyzed (Participants) | 20
participants | 20

4. Secondary Outcome: Fluoroscopy Time
Description: As recorded by an X-ray system utilized during the procedure.
Time Frame: Procedure
Population: Procedure time for subjects measured from the insertion of the hemostasis sheath until the removal of the guide catheter.
Measure: Mean (Standard Error); unit: min
Groups:
- Fluoroscopy and/or X-ray Time: As recorded by an X-ray system utilized during the procedure.
Arm/Group | Fluoroscopy and/or X-ray Time
Number analyzed (Participants) | 20
min | 6.8 (3.4)

5. Secondary Outcome: Contrast Volume
Description: Total amount of contrast used during CorPath procedure.
Time Frame: Procedure
Population: Total amount of contrast used during CorPath procedure for subjects.
Measure: Mean (Standard Error); unit: ml
Groups:
- Contrast Fluid Volume: Total amount of contrast used during CorPath procedure.
Arm/Group | Contrast Fluid Volume
Number analyzed (Participants) | 20
ml | 73.3 (9.2)

6. Secondary Outcome: Total Procedure Time
Description: Defined as the time measured from the insertion of the hemostasis sheath until procedure complete (guide catheter removed).
Time Frame: Procedure
Population: Total procedure time for subjects.
Measure: Mean (Standard Deviation); unit: min
Groups:
- Overall Procedure Time: Defined as the time measured from the insertion of the hemostasis sheath until procedure complete (guide catheter removed).
Arm/Group | Overall Procedure Time
Number analyzed (Participants) | 20
min | 45.5 (6.2)

7. Secondary Outcome: Interventional Procedure Time
Description: Defined as the time measured from the insertion of the guide catheter until the removal of the guide catheter.
Time Frame: Procedure
Population: Interventional procedure time for subjects.
Measure: Mean (Standard Deviation); unit: min
Groups:
- PVI Procedure Time: Defined as the time measured from the insertion of the guide catheter until the removal of the guide catheter.
Arm/Group | PVI Procedure Time
Number analyzed (Participants) | 20
min | 23.4 (14.0)

ADVERSE EVENTS:
Time Frame: All subjects will be followed post-CorPath procedure through 24 hours or hospital discharge, whichever occurs first.
Arm/Group | Device-related Periprocedural Event
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This study represents a single high-volume tertiary care center experience and the results need to be replicated by multiple users to show the general applicability of these findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No